CLINICAL TRIAL: NCT05561959
Title: Efficacy of Phonophoresis With Topical Glyceryl Trinitrate in Treatment of Non-insertional Achilles Tendinopathy: a Randomized Controlled Trial
Brief Title: Efficacy of Phonophoresis With Topical Glyceryl Trinitrate in Treatment of Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, lecturer of physical therapy Basic Science department faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012
Record Dates: First submitted 2022-09-19; First posted 2022-09-30 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Non Insertional Achilles Tendinopathy
Keywords: Achilles tendinopathy; phonophoresis; topical glyceryl trinitrate

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phonophoresis Group (Experimental): Phonophoresis with topical glyceryl trinitrate traditional therapy three times a week for four week
  Interventions: Other: topical glyceryl trinitrate gel
- Eccentric exercises Group (Active Comparator): eccentric exercises three times a week for four weeks
  Interventions: Other: Eccentric exercises

INTERVENTIONS:
Other: topical glyceryl trinitrate gel — topical nitroglycerin medication were treated with 1 gr nitroglycerin 2% gel
  Arms: Phonophoresis Group
Other: Eccentric exercises — stretching exercises of the gastrocnemius (straight leg) and soleus (bended knee).
  Arms: Eccentric exercises Group

SUMMARY:
The aim of study is to investigate the effect of Phonophoresis with topical glyceryl trinitrate versus traditional treatment in in patients with non-insertional Achilles tendinopathy.

DETAILED DESCRIPTION:
Pain in the Achilles tendon is quite common in individuals who participate in sports It is also common, however, in nonathletic individuals, particularly in persons of middle age who are of heavier weight Treating this condition can be very challenging. It is seen most commonly in the mid-portion of the tendon. The pathologic changes that occur to an Achilles tendon under repetitive stress will initially be a disruption of collagen fibers that have been unable to adapt to the persistent demand. This results in a cascade of events that, if left unchecked, will ultimately lead to significant pain and dysfunction. Repetitive loading leads to tendon degeneration, manifested as loss of normal collagen patterns and replacement of normal tissue with disorganized arrays of collagen and proliferative extracellular matrix. The tendon becomes infiltrated with mucoid material, calcification, fibrocartilage, and lipid droplets.

Historically, one of the most well-established exercise regimens for Achilles tendinopathy is eccentric strength training. Eccentric exercise has been shown to improve tendon structure, which historically was considered a mechanism for improvement in some persons with Achilles tendinopathy.

Nitric oxide is a small-free radical generated by a family of enzymes, the nitric oxide synthases. In a series of experiments performed over the last 15 years, nitric oxide played a crucial beneficial role in restoring tendon function. Oxygen free radicals, in the correct dose, stimulated fibroblast proliferation. Nitric oxide can enhance tendon healing. Nitric oxide is 1 of the 10 smallest molecules. Its size and its high reactivity allow it to travel across nearly all biologic structures and to readily react with other atoms or molecules to effect a change.

so the aim of our study to compare between Phonophoresis with topical glyceryl trinitrate and eccentric strength training in treatment of Achilles tendinopathy

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-50 years old
2. The diagnosis was based on pain located in the Achilles tendon for at least 3 months.
3. Pain in the Achilles tendon area with distinct tenderness of the tendon 2 to 6 cm above the Achilles tendon insertion on the calcaneus
4. Ultrasonographic changes defined as local thickening of the symptomatic tendon, irregular tendon structure and fiber orientation, and separated tendon fibers or a globally more than 2 mm thicker tendon on the sick side
5. Diffuse pain in the posterior region of the ankle with local tenderness of the Achilles tendon and ultrasonographic changes.

Exclusion Criteria:

1. Symptoms of <3 months, previous surgery, previous ankle dislocation, distal neurology, steroid injections in last 3 month, pregnancy, and contraindication to GTN
2. Treatment of achillodynia with stretching or eccentric training for more than 2 weeks within the last 2 years
3. Other injuries in the lower extremity or the knee, which by the examining doctor was evaluated to influence the evaluation of symptoms or the ability to perform the training program
4. Acute symptoms with ultrasonographic changes consistent with a partial rupture of the tendon

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
the change in thickness of Achilles tendon | at first week and after 12 week of treatment
  measured by Ultrasonography.
the change in Pain in patients with non-insertional Achilles tendinopathy. | at first week and after 12 week of treatment
  measured by Visual Analog Scale
the change in Functional performance | at first week and after 12 week of treatment
  measured by vertical countermovement jump test.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No